CLINICAL TRIAL: NCT04661267
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Regenexx Stem Cell Support Formula
Brief Title: Randomized Trial of Regenexx Stem Cell Support Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RGX2020-RCT02
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement formula (Experimental): Patients randomized to the experimental group will receive daily 1-ounce doses of stem cell support formula for 60 days. Patients will complete patient-reported outcome questionnaires at 1 month and 2 months.
  Interventions: Dietary Supplement: Stem Cell Support Formula
- Placebo formula (Placebo Comparator): Patients randomized to the control group will receive a daily 1-ounce doses of placebo stem cell support formula for 60 days. Patients will complete patient-reported outcome questionnaires at 1 month and 2 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Stem Cell Support Formula — This liquid supplement contains the following ingredients: chondroitin sulfate, glucosamine sulfate, vitamin C (ascorbic acid), curcumin and Bioperine®, resveratrol, L-carnosine, bitter melon, and vitamin D.
  Arms: Supplement formula
Dietary Supplement: Placebo — The placebo comparator will look and taste similar without the active ingredients of the Stem Cell Support Formula.
  Arms: Placebo formula

SUMMARY:
Regenexx, LLC developed a nutritional supplement formula containing many components related to supporting healthy joints This oral, liquid supplement is intended to help improve joint and cartilage health while also increasing their joint function. The goal of this study is to measure changes in joint health and function for patients with knee OA taking this supplement for 2 months.

DETAILED DESCRIPTION:
The study design is a double-blind, randomized, placebo-controlled multicenter study. Liquid Regenexx Stem Cell Support Formula compared to placebo control administered via oral application for 2 months to determine effect on knee function and pain in patients with knee OA.

Treatment group: Forty patients randomized to the treatment group will receive daily doses of stem cell support formula for 60 days. Patients will complete patient-reported outcome questionnaires at 1 month and 2 months.

Control group: Forty patients randomized to the control group will receive a daily doses of placebo stem cell support formula for 60 days. Patients will complete patient-reported outcome questionnaires at 1 month and 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signature of the IRB approved Informed Consent
2. Unilateral or bilateral osteoarthritic male or female ages 18-80
3. Pain, swelling, and/or functional disability in the affected knee consistent with osteoarthritis in the knee joint
4. Physical examination consistent with osteoarthritis in knee joint
5. Kellgren-Lawrence grade 2 or 3 knee osteoarthritis and/or diagnostic MRI imaging of the affected knee showing osteoarthritis (i.e. chondral loss, fissuring, defect, bone marrow lesion, meniscus tear, synovial thickening, etc.)
6. Minimum of 3/10 on NPS approximately 3 days per week
7. Is independent, ambulatory, and can comply with all post-operative evaluations and visits

   Exclusion Criteria:
8. Previously taken the Regenexx Stem Cell Support Formula
9. Receiving active knee treatment or any knee injections of any type within 3 months prior to the study (steroids, biologics, etc)
10. Knee surgery within 6 months prior to the study
11. Currently taking or history of taking products that contain curcuminoid extract within the last 2 weeks
12. Dependent on NSAIDs or acetaminophen for exercise or daily activities
13. Currently taking or previously taken fish oil in the last 2 weeks
14. Currently taking or previously taking MSM or glucosamine in the last 2 weeks
15. Diabetic
16. Inflammatory or auto-immune based joint diseases or other lower extremity pathology (e.g., rheumatoid arthritis, systemic lupus erythematosus, psoriatic arthritis, polymyalgia, polymyositis, gout pseudogout)
17. Quinolone or statin-induced myopathy/tendinopathy
18. Severe neurogenic inflammation of the cutaneous nerves about the knee or thigh
19. Contraindications for MRI
20. Condition represents a worker's compensation case
21. Currently involved in a health-related litigation procedure
22. Is pregnant or breastfeeding
23. Currently taking immunosuppressive medication
24. Allergy or intolerance to study medication
25. Use of chronic opioid
26. Documented history of drug abuse within six months of treatment
27. Blood clotting disorder, taking an anticoagulant or history of cardiovascular disease
28. Has asthma
29. History of prostate cancer

29) Any other condition, that in the opinion of the investigator, that would preclude the patient from enrollment including current supplement use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Lower Extremity Function Scale (LEFS) change from baseline | Change from baseline to 2 months
  The difference between groups of the within patient mean change from baseline to 2 months.
Minimal Clinically Important Difference (MCID) for LEFS | 2 months
  Percentage of patients meeting the MCID for LEFS at 2 months

SECONDARY OUTCOMES:
Lower Extremity Function Scale (LEFS) change from baseline | Change from baseline to 1 month
  The difference between groups of the within patient mean change from baseline to 1 month.
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation change from baseline | Change from baseline to 2 months
  The difference between groups of the within patient mean change from baseline to 2 months
International Knee Documentation Committee (IKDC) Subjective Knee Evaluation change from baseline | Change from baseline to 1 months
  The difference between groups of the within patient mean change from baseline to 1 months
Minimal Clinically Important Difference (MCID) for IKDC | 2 months
  Percentage of patients meeting the MCID for IKDC at 2 months
Numeric Pain Score (NPS) change from baseline | Change from baseline to 1 months
  The difference between groups of the within patient mean change from baseline to 1 month.
Numeric Pain Score (NPS) change from baseline | Change from baseline to 2 months
  The difference between groups of the within patient mean change from baseline to 2 months.
Minimal Clinically Important Difference (MCID) for NPS | 2 months
  Percentage of patients meeting the MCID for NPS at 2 months
Single Assessment Numeric Evaluation (SANE)-modified | 1 month
  The difference between groups for mean improvement scores at 1 month
Single Assessment Numeric Evaluation (SANE)-modified | 2 months
  The difference between groups for mean improvement scores at 2 months
Adverse events | Thru 2 months
  Any complication or adverse event reported
Additional medications or treatments | Thru 2 months
  Any additional treatments or medications

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Regenexx, LLC and Centeno-Schultz Clinic
Locations (2):
- United States (2):
  - Centeno-Schultz Clinic, Broomfield, Colorado
  - Centeno-Schultz Clinic, Lone Tree, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Someya A, Ikegami T, Sakamoto K, Nagaoka I. Glucosamine Downregulates the IL-1beta-Induced Expression of Proinflammatory Cytokine Genes in Human Synovial MH7A Cells by O-GlcNAc Modification-Dependent and -Independent Mechanisms. PLoS One. 2016 Oct 24;11(10):e0165158. doi: 10.1371/journal.pone.0165158. eCollection 2016. PMID 27776166
- [Background] Jerosch J. Effects of Glucosamine and Chondroitin Sulfate on Cartilage Metabolism in OA: Outlook on Other Nutrient Partners Especially Omega-3 Fatty Acids. Int J Rheumatol. 2011;2011:969012. doi: 10.1155/2011/969012. Epub 2011 Aug 2. PMID 21826146
- [Background] Du CB, Liu JW, Su W, Ren YH, Wei DZ. The protective effect of ascorbic acid derivative on PC12 cells: involvement of its ROS scavenging ability. Life Sci. 2003 Dec 26;74(6):771-80. doi: 10.1016/j.lfs.2003.07.014. PMID 14654169
- [Background] D'Aniello C, Cermola F, Patriarca EJ, Minchiotti G. Vitamin C in Stem Cell Biology: Impact on Extracellular Matrix Homeostasis and Epigenetics. Stem Cells Int. 2017;2017:8936156. doi: 10.1155/2017/8936156. Epub 2017 Apr 20. PMID 28512473
- [Background] Larasati YA, Yoneda-Kato N, Nakamae I, Yokoyama T, Meiyanto E, Kato JY. Curcumin targets multiple enzymes involved in the ROS metabolic pathway to suppress tumor cell growth. Sci Rep. 2018 Feb 1;8(1):2039. doi: 10.1038/s41598-018-20179-6. PMID 29391517
- [Background] Leonard SS, Xia C, Jiang BH, Stinefelt B, Klandorf H, Harris GK, Shi X. Resveratrol scavenges reactive oxygen species and effects radical-induced cellular responses. Biochem Biophys Res Commun. 2003 Oct 3;309(4):1017-26. doi: 10.1016/j.bbrc.2003.08.105. PMID 13679076
- [Background] Prasad S, Tyagi AK, Aggarwal BB. Recent developments in delivery, bioavailability, absorption and metabolism of curcumin: the golden pigment from golden spice. Cancer Res Treat. 2014 Jan;46(1):2-18. doi: 10.4143/crt.2014.46.1.2. Epub 2014 Jan 15. PMID 24520218
- [Background] Prokopieva VD, Yarygina EG, Bokhan NA, Ivanova SA. Use of Carnosine for Oxidative Stress Reduction in Different Pathologies. Oxid Med Cell Longev. 2016;2016:2939087. doi: 10.1155/2016/2939087. Epub 2016 Jan 24. PMID 26904160
- [Background] Dandawate PR, Subramaniam D, Padhye SB, Anant S. Bitter melon: a panacea for inflammation and cancer. Chin J Nat Med. 2016 Feb;14(2):81-100. doi: 10.1016/S1875-5364(16)60002-X. PMID 26968675